CLINICAL TRIAL: NCT02763293
Title: Soft Ostheopathic Techniques Improve the Quality of Life in Patients With Crohn's Disease. A Randomized Controlled Trial.
Brief Title: Osteopathy Non-manipulative in Patients With Crohn's Disease.
Acronym: ONManCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, University of Valencia
Allocation: Non-Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ID013
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Crohn´s Disease
Keywords: pain; effectiveness; manual therapy
MeSH Terms: conditions — Crohn Disease; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy (Experimental): Cranial therapy (CT). Neuro-lymphatic reflexes treatment (NL) Viscerosomatic reflexes (VR) Induction myofascial Visceral osteopathic therapy (VOT)
  Interventions: Other: Manual Therapy
- Control Group (No Intervention): Patients only came to make assessments, without receiving any treatment.

INTERVENTIONS:
Other: Manual Therapy — Non-manipulative treatment osteopathic techniques combined direct and indirect soft appropriate in patients with Crohn's disease
  Arms: Manual Therapy

SUMMARY:
Crohn's disease (CD) is an inflammatory bowel disease with a high prevalence. Its etiology is unknown and is considered a multifactorial disease. It is known that the existence of a genetic factor, industrialization and development of the country and environmental factors have great influence on the appearance of intestinal pathology (the Val; Buderus; Molodecky). CD is a chronic inflammatory bowel disease localized throughout the course of the digestive tract (oral-anal). The aim of this study is to evaluate the effect of a treatment program combining technical nonmanipulative appropriate in affected patients (CD) to increase the overall quality of life and related EC, lower abdominal pain direct and indirect osteopathic soft, observe the sense of change after treatment, and psychological aspects.

DETAILED DESCRIPTION:
All of the participants were recruited, in a non-probabilistic way, from the Valencian Association of Enfermos de Crohn y Colitis Ulcerosa (ACCU) The participants were allocated to two different groups depending on their possibility of participation in the therapeutic sessions. The group that received the therapy was called experimental group (EG) and the group, who did not, control group (CG). The participants were allocated independently of their disease status (outbreak or remission).

An experimental study carried out during a period of four weeks in order to explore the effect of the specific treatment on the following outcomes: global quality of life, quality of life in CD and pain.

The participants, in the EG were treated in three sessions, that lasted 45 minutes, during the study duration (1 session each 9-10 days). The physiotherapist who applied the treatment had an extensive experience in manual therapy.

Both groups come to laboratory two times for the assessment, one at the beginning of the study and the other one at the end. In each session several questionnaires were administered by a physiotherapist who was blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with active CD of at least one year of evolution, aged between 18 and 65, with a presence of abdominal pain, receiving conservative or surgical treatment (after 6 months after surgery and absence of diverting ileostomy) were included. Once they expressed their interest in taking part of the study, potential participants underwent an examination by a specialist of the association to confirm the diagnosis of CD.

Exclusion Criteria:

* Conversely, patients with non-specific inflammatory bowel, abdominal tenderness, infection, ischaemia, physical damage, or specific immunologic sensitivity or pregnancy be excluded of this study were discarded for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain. | 4 weeks
  by a horizontal line 10 cm in length (0 = no pain to 10 = maximum pain).

SECONDARY OUTCOMES:
Global Quality Of Life | 4 weeks
  Functional Assessment of Cancer Therapy- General (Versión 4- FACT-G)
Quality Of Life in CD | 4 weeks
  Inflammatory Bowel Disease Quality Of Life-32 (IBDQ-32)
Index of Crohn's disease activity | 4 weeks
  By the Harvey-Bradshaw Index (HBI)
Existence of anxiety and depression | 4 weeks
  by Goldberg Anxiety and Depression Scale
Anxiety and Depression | 4 weeks
  Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Espí, Principal Investigator — Faculty of Physiotherapy
Locations (1):
- Faculty of Physiotherapy, Valencia, Spain

REFERENCES:
- [Result] Piche T, Pishvaie D, Tirouvaziam D, Filippi J, Dainese R, Tonohouhan M, DeGalleani L, Nebot-Vivinus MH, Payrouse JL, Hebuterne X. Osteopathy decreases the severity of IBS-like symptoms associated with Crohn's disease in patients in remission. Eur J Gastroenterol Hepatol. 2014 Dec;26(12):1392-8. doi: 10.1097/MEG.0000000000000219. PMID 25357218
- [Result] Florance BM, Frin G, Dainese R, Nebot-Vivinus MH, Marine Barjoan E, Marjoux S, Laurens JP, Payrouse JL, Hebuterne X, Piche T. Osteopathy improves the severity of irritable bowel syndrome: a pilot randomized sham-controlled study. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):944-9. doi: 10.1097/MEG.0b013e3283543eb7. PMID 22546751